CLINICAL TRIAL: NCT05614895
Title: A Multicenter, Single-Dose, Uncontrolled, Open-label, One Group Study to Investigate the Pharmacokinetics of RO7223280 in Critically Ill Patients With Bacterial Infections
Brief Title: A Study to Investigate the Pharmacokinetics of RO7223280 in Critically Ill Participants With Bacterial Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP43949; 2022-000456-11 (EudraCT Number); ISRCTN21709018 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2022-11-10; First posted 2022-11-14 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Bacteremia participants without pneumonia and who are not mechanically ventilated at screening will be enrolled in this cohort. Participants will receive RO7223280 on Day 1.
  Interventions: Drug: RO7223280
- Cohort 2 (Experimental): Participants with hospital-acquired bacterial pneumonia (HABP) and who are not mechanically ventilated at screening will be enrolled in this cohort. Participants will receive RO7223280 on Day 1.
  Interventions: Drug: RO7223280
- Cohort 3 (Experimental): Participants with mechanical ventilation at screening will be enrolled in this cohort. Participants will receive RO7223280 on Day 1.
  Interventions: Drug: RO7223280
- Cohort 4 (Experimental): Participants with mechanical ventilation who have a bronchoalveolar lavage (BAL) planned as a part of routine practice will be enrolled in this cohort. Participants will receive RO7223280 on Day 1.
  Interventions: Drug: RO7223280

INTERVENTIONS:
Drug: RO7223280 — Participants will receive RO7223280, 600 mg, IV infusion for 1 hour on Day 1.
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: RO7223280 — Participants will receive RO7223280, 400 mg, IV infusion for 1 hour on Day 1.
  Arms: Cohort 4

SUMMARY:
The main aim of the study is to investigate the plasma pharmacokinetics (PK) and safety of intravenous (IV) administration of a single dose of 400 milligrams (mg) or 600 mg RO7223280 in critically ill participants with bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* Illness requiring treatment in an intensive care unit (ICU) at the time of enrolment
* Ongoing clinical syndrome meeting at least one of the following criteria:

  1. HABP: bacterial pneumonia diagnosed after more than 48 hours of hospitalization or within 7 days after a hospital discharge
  2. Ventilator-associated bacterial pneumonia (VABP): bacterial pneumonia diagnosed after more than 48 hours of mechanical ventilation or within 72 hours after weaning
  3. Bacteremia confirmed by the presence of a bacterial pathogen in a blood culture drawn within 7 days prior to dosing and with the defined focus of infection.
  4. For Cohort 4 only: mechanically ventilated participants who have a BAL procedure planned as part of routine practice for a day that can function as Day 1.

Exclusion Criteria:

* Ongoing documented catheter-related bacteraemia as the sole ongoing infection
* Major surgery within 48 hours prior to dosing or major surgery expected within 48 hours after the start of the infusion
* Known chronic severe hepatic impairment (Child-Pugh class C). Note: acute severe hepatic impairment is not exclusionary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of RO7223280 | Cohort 1-3: From Day 1 up to Day 3; Cohort 4: From Day 1 up to Day 5

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Cohort 1-3: From Day 1 up to Day 4; Cohort 4: From Day 1 up to Day 5
Percentage of Participants With Serious Adverse Events (SAEs) | Cohort 1-3: From Day 1 up to Day 4; Cohort 4: From Day 1 up to Day 5
Percentage of Participants Who Died Due to Any Cause | Cohort 1-3: From Day 1 up to Day 4; Cohort 4: From Day 1 up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (5):
  - Infectious Disease Associates, Sarasota, Florida
  - University of Louisville Physicians, Louisville, Kentucky
  - Beaumont Hospital; Royal Oak Pharmacy, Royal Oak, Michigan
  - East Carolina University (ECU) Physicians - Infectious Disease Clinic - Greenville, Greenville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
- France (5):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpitaux Universitaires de strasbourg - hôpital civil, Strasbourg
- Israel (3):
  - Hadassah Ein Karem Hospital, Jerusalem
  - The Chaim Sheba Medical Center; Multiple Sclerosis Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- ARENSIA Phase 1 Unit- Spitalul Clinic Republican Location, Chisinau, Moldova
- South Korea (2):
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Asan Medical Center., Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical -trials/data-sharing/).